CLINICAL TRIAL: NCT05381389
Title: Onset and Recovery of Ultrasound Guided Out-of-plane Versus In-plane Interscalene Block in Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada M.Samir, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU R59/2018
Record Dates: First submitted 2022-05-12; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group In-plane approach: (Active Comparator): An in-plane approach was used for the interscalene block. The needle was brought in the same plane as the probe at a shallow angle to the skin, some distance away from the edge of the probe in a lateral to medial direction so that the whole length of the needle can be visualized. After negative aspiration and assurance that high resistance to injection was absent, the LA was injected in a 5 ml increment below the lower root, between the 3 roots and above the upper root.
  Interventions: Drug: Bupivacaine Hydrochloride in-plane approach for the interscalene block
- Group Out-of-plane approach (Active Comparator): An out-of-plane approach was used for the interscalene block. The needle was inserted cranial to the probe and after negative aspiration and assurance that high resistance to injection was absent, the LA was injected in a 10 ml increment; lateral and medial to the nerve roots. The needle appeared as a bright dot on the screen and by tilting the probe, the tip was identified as the point where further tilting leads to no longer visualization of the bright dot on the screen.
  Interventions: Drug: Bupivacaine Hydrochloride out of-plane approach for the interscalene block

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride in-plane approach for the interscalene block — 20 ml of 0.5% bupivacaine added to them 50 μg adrenaline in a concentration of 1:400,000, were prepared by an assistant immediately before administration and injected in an in-plane approach to the brachial plexues
  Arms: Group In-plane approach:
Drug: Bupivacaine Hydrochloride out of-plane approach for the interscalene block — 20 ml of 0.5% bupivacaine added to them 50 μg adrenaline in a concentration of 1:400,000, were prepared by an assistant immediately before administration and injected in an out of-plane approach to the brachial plexues
  Arms: Group Out-of-plane approach

SUMMARY:
The aim of this study was to assess the out-of-plane versus the in-plane approaches for the interscalene brachial plexus block; as regards the performance time, the onset, the progression and the recovery of sensory block, the onset and progression of the motor block as well as, the postoperative pain score and the duration of analgesia for arthroscopic shoulder surgery. A total of 60 patients of American Society of Anesthesiologists (ASA) physical status I-II were randomly divided to receive either the in-plane approach (Group I), or the out-of-plane approach (Group O).

DETAILED DESCRIPTION:
60 patients of ASA physical status I - II, greater than or equal to 30 years old and smaller than or equal to 60 years old, scheduled to undergo arthroscopic shoulder surgery in the lateral position; under ultrasound -guided interscalene brachial plexus block (ISPB) in this randomized study at Ain-Shams University Hospitals. On arriving to the operating theater, patients had an 18G intravenous cannula inserted in the non-operative upper limb side. All patients received; 0.05 mg/kg IV midazolam hydrochloride and 30 mg pethidine. Intraoperative basic monitors were applied using 5-leads ECG, pulse oximetry, non-invasive blood pressure (NIBP) and capnography (sample tube inserted under the O2 mask).A simple O2 mask at a flow of 6L/min was applied. Infusion of Ringer's solution was then started at a rate of 5mL/kg/h throughout the surgery. Patients were placed in the supine position with their heads rotated towards the non-operative side. Iodine solution was used as an antiseptic on the operative neck side and then the patient head, neck and chest were draped. Local infiltration of the skin at the point of needle insertion was carried out with 2 ml lidocaine hydrochloride 1%, then a sterile 50-mm 22-G insulated needle was used for performance of the block.The ultrasound with a high frequency linear transducer was used, with the depth setting of 2-4 cm. Distal to proximal (Trace back) approach was used; the supraclavicular fossa was scanned first to identify the subclavian artery as it passes over the first rib; by placing the probe against the clavicle and scanning in a caudate direction. The brachial plexus was easily identified as bunch of grapes supero-lateral to the artery. The plexus was followed medially and cephalad along its course by keeping the nerves in the center of the screen, to identify the brachial plexus roots between the anterior and the middle scalene muscles at the level of the sixth cervical vertebra deep to the sternocleidomastoid muscle.

Patients were then divided into 2 equal groups of 30 patients each:

Group I: An in-plane approach was used for the interscalene block. The needle was brought in the same plane as the probe at a shallow angle to the skin, some distance away from the edge of the probe in a lateral to medial direction so that the whole length of the needle can be visualized. After negative aspiration and assurance that high resistance to injection was absent, the LA was injected in a 5 ml increment below the lower root, between the 3 roots and above the upper root.

Group O: An out-of-plane approach was used for the interscalene block. The needle was inserted cranial to the probe and after negative aspiration and assurance that high resistance to injection was absent, the LA was injected in a 10 ml increment; lateral and medial to the nerve roots. The needle appeared as a bright dot on the screen and by tilting the probe, the tip was identified as the point where further tilting leads to no longer visualization of the bright dot on the screen.

After completion of the LA administration, the time was recorded as a baseline for the time interval. The assistant who recorded the data was blind to the patient groups. The sensory block was assessed by a pin-prick test using a 3-point scale. The motor block was assessed according to the shoulder, arm and fingers movement using a 3-point scale. Postoperative pain was measured at rest using the VAS score

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I - II
* scheduled to undergo arthroscopic shoulder surgery in the lateral position

Exclusion Criteria:

* body mass index ≥ 35 kg/m2 body surface area
* anticipated difficult airway
* infection at the injection site
* known LA allergy,
* contralateral phrenic nerve dysfunction
* history of cardiac disease
* history of hepatic disease
* history of renal disease
* coagulopathy
* chronic obstructive pulmonary disease
* neuropathy involving the brachial plexus.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
The onset of sensory block (time to C5 block) | 30 minutes
  defined as the period between the completion of the LA administration and the loss of sensation to pin prick in C5 dermatome performed every 1 minute

SECONDARY OUTCOMES:
The procedure time | 20 minutes
  time from the skin infiltration by the lidocaine till removal of the stimulating needle from the skin
Progression of sensory block | over the first 20 minutes of LA injection
  performed by pin prick every 5 minutes in C6, C7, C8 and T1 dermatomes
The onset of motor block | 30 minutes
  the period between the completion of LA administration till lack of movement of the shoulder, arm and fingers muscles assessed every 1 minute.
The progression of motor block | over the first 20 minutes of LA injection
  in the shoulder, arm and fingers muscles assessed every 5 minutes
The duration of motor block | 24 hours
  the period between the onset of motor block till complete recovery of motor function
Postoperative pain score | 24 hours
  Intensity of pain was monitored at rest
The duration of analgesia | 24 hours
  the time interval between the onset of sensory block until the first call for analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No